CLINICAL TRIAL: NCT03598400
Title: Can High Intensity Interval Training Reduce Fear of Hypoglycaemia and Improve Glycaemic Control in People With Type 1 Diabetes?
Brief Title: HIT on Hypoglycemic Risk in Type 1 Diabetes (T1D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Society for Endocrinology (Other); Royal Liverpool University Hospital (Other Government); University of Birmingham (Other); University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: T1D1
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-02

CONDITIONS: Type1diabetes
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will continue with their habitual lifestyle but perform no exercise for 2 weeks
- Moderate intensity continous training (Active Comparator): Participants will complete moderate intensity continous training during a 2 week intervention period
  Interventions: Behavioral: moderate intensity continous training
- high intensity interval training (Experimental): Participants will complete high intensity interval training during a 2 week intervention period
  Interventions: Behavioral: high intensity interval training

INTERVENTIONS:
Behavioral: high intensity interval training — Participants will complete 6 sessions of high intensity interval training during a 2 week intervention period. The programme involves repeated 1 minute bouts of simple on the spot movements interspersed with 1 minute of rest.
  Arms: high intensity interval training
Behavioral: moderate intensity continous training — Participants will complete 6 sessions of moderate intensity continous training during a 2 week intervention period. Participants will be asked to complete 30 minutes of continuous exercise.
  Arms: Moderate intensity continous training

SUMMARY:
There is clear evidence that regular exercise improves wellbeing and reduces the risk of diabetes related complications in people with type 1 diabetes. However, many people with type 1 diabetes do not exercise regularly. The primary reason for this is fear of hypoglycaemia and loss of glycaemic control associated with exercise. This loss of glycaemic control is associated with traditional moderate intensity continous aerobic exercise advocated in the guidelines for exercise in people with type 1 diabetes. Recent work (unpublished) from our lab suggests high intensity interval training (HIT) may reduce the risk of hypoglycaemia in people with type 1 diabetes, however stronger evidence is needed before firm conclusions can be drawn.

Therefore, the aim of this study is to determine the effects of HIT on glycaemic control in people with type 1 diabetes compared to no exercise and traditional moderate intensity continous exercise.

24 people with type 1 diabetes will be recruited to complete a randomised counterbalanced cross over study comparing 3x 2-week interventions periods. During these intervention periods participant will maintain their habitual lifestyle but complete either no exercise (control), traditional moderate intensity continous exercise or high intensity interval training. Throughout the intervention periods participants glycaemic control will be monitored using a flash glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis more than 6 months ago (to ensure participants are out of the honeymoon period),
* Using a basal bolus insulin regime or insulin pump therapy
* BMI ≤ 32 kg.m-2

Exclusion Criteria:

* Pregnancy (or planning pregnancy)
* Disability preventing participation in an exercise regime
* Angina
* Autonomic neuropathy
* Medication that affects heart rate (this will affect estimation of fitness)
* Major surgery planned within 6 weeks of study
* Uncontrolled blood pressure
* Significant history of hyperglycaemia
* History of severe hypoglycaemia requiring third party assistance within the last 3 months
* Severe non-proliferative and unstable proliferative retinopathy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Severe hypoglycaemia | 2 weeks
  Number of severe hypoglycaemic events (<3mmol/l) during the 2 week intervention period

SECONDARY OUTCOMES:
Mean glucose | 2 weeks
  mean glucose level over 2 week recording period
% of time in level 2 hypoglycaemia (<3.0mmol/L) | 2 weeks
  % of time in level 2 hypoglycaemia (<3.0mmol/L) over 2 week recording period
% of time in level 1 hypoglycaemia (3.0-3.9mmol/L) | 2 weeks
  % of time in level 1 hypoglycaemia (3.0-3.9mmol/L) over 2 week recording period
% of time in target range (3.9-10.0mmol/L) | 2 weeks
  % of time in target range (3.9-10.0mmol/L) over 2 week recording period
% of time in level 1 hyperglycaemia (10.0-13.9mmol/L) | 2 weeks
  % of time in level 1 hyperglycaemia (10.0-13.9mmol/L) over 2 week recording period
% of time in level 2 hyperglycaemia (>13.9mmol/L) | 2 weeks
  % of time in level 2 hyperglycaemia (>13.9mmol/L) over 2 week recording period
glycaemic variability (coefficient of variation and Standard Deviation) | 2 weeks
  glycaemic variability over 2 week recording period
area under the curve of episodes of hypoglycaemia and hyperglycaemia | 2 weeks
  area under the curve of episodes of hypoglycaemia and hyperglycaemia 2 week recording period

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared outside the research team. Anonymised group data will be presented in research articles and presentations